CLINICAL TRIAL: NCT00815945
Title: Phase II Study Evaluating PegLiposomal Doxorubicin (PLD) and Carboplatin Combination Chemotherapy in Gynecological Sarcomas and Mixed Epithelial-Mesenchymal Tumors
Brief Title: Multicenter Trial With PegLiposomal Doxorubicin and Carboplatin Combination Chemotherapy in Gynecological Sarcomas and Mixed Epithelial-Mesenchymal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO-GYN 7
Record Dates: First submitted 2008-12-30; First posted 2008-12-31 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2014-03

CONDITIONS: Mesenchymal Tumor; Carcinosarcoma; Leiomyosarcoma
Keywords: leiomyosarcoma; carcinosarcoma; mixed epithelial mesenchymal tumor; endometrial stroma sarcomas; Müllerian mixed tumors; carcinosarcoma of the uterus; mesenchymal tumors of the ovary or uterus; mixed epithelial mesenchymal tumors of the ovary or uterus
MeSH Terms: conditions — Carcinosarcoma; Leiomyosarcoma | interventions — liposomal doxorubicin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PegLiposomal Doxorubicin + Carboplatin (Experimental): Subjects will receive PegLiposomal Doxorubicin (40mg/m²) and Carboplatin (AUC6) every 28 days. Treatment period up to 6 months (therapy can be continued in case of tumor response and benefit for the patient)
  Interventions: Drug: PegLiposomal Doxorubicin; Drug: Carboplatin

INTERVENTIONS:
Drug: PegLiposomal Doxorubicin — PegLiposomal Doxorubicin, intravenous, 40mg/m², every 28 days for up to 6 months
  Other Names: Caelyx
Drug: Carboplatin — Carboplatin, intravenous, AUC 6, every 28 days for up to 6 months

SUMMARY:
Uterine sarcomas account for less than 5% of all carcinomas of the uterine corpus. The prognosis of these patients is extremely limited. Recurrence rates of 50-60% are reported even for early-stage disease (FIGO I/II). Median overall survival is below 12 months in patients with advanced or metastatic disease.

Ovarian carcinosarcoma is extremely rare among ovarian malignancies (< 2%). That is why there is insufficient data as a basis for establishing a gold standard. As a result, these cases tend to be treated in the same way as uterine sarcomas or epithelial ovarian malignancies in clinical practice.

On the basis of data published to date on the treatment of mixed mesenchymal-epithelial tumors, it is clear that the treatments commonly used to date have limited activity while producing clinically relevant toxicity. The regimes verified so far (Cisplatin / Ifosfamide, Ifosfamide/Paclitaxel and Gemcitabine/Docetaxel) exhibit a considerable side effect spectrum and are only rarely feasible on clinical everyday life conditions, so e. g. the rate of withdrawals due to toxicity was in a study collective of selected females treated with the last combination at 40 %. The physician has to check in every individual case if one of the above mentioned combinations is feasible. The search for alternative effective and better tolerated treatment options is essential. The toxicity data on the carboplatin-PLD combination are known, and efficacy has been identified in small cohorts.

The objective of this study is to explore the efficacy of combination PLD-carboplatin treatment in a larger patient population.

DETAILED DESCRIPTION:
This study in patients with mesenchymal or mixed epithelial mesenchymal tumors of the ovary or uterus is designed as a prospective single-arm, open - label, multicenter phase II study to evaluate the efficacy of PegLiposomal Doxorubicin and Carboplatin combination chemotherapy.

40 patients will be recruited to receive PegLiposomal Doxorubicin (PLD) in a continuous i. v. infusion of at least 60 minutes at a dose of 40 mg/m2 on Day 1, followed by a 30-minute i. v. carboplatin infusion according to AUC 6 (formula devised by Calvert et al).

Patients will get outpatients treatment. At screening the patients' eligibility will be assessed, their baseline and demographic characteristics obtained, and baseline values for the effect variables collected. Patients with measurable lesions, non-measurable lesions or histological documentation will be included into this trial. Measurable lesion and non-measurable lesions will be documented by x-ray, ultrasound, computed tomography or MRI.

The patients' safety will be monitored during therapy until recovery of toxicities.

In patients with measurable lesions at baseline, the (post)-treatment values for effect according to the RECIST criteria will be collected as shown in table 6. CR, PR and SD have to be confirmed by a repeat measurement after an interval of at least four weeks.

Follow-up is scheduled every three months during the first two years after the end of treatment.

As from year 3 the follow-up takes place outside the study in the context of general aftercare.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented mesenchymal or mixed epithelial-mesenchymal tumor of the ovary or uterus
* Patients with a primary diagnosis of FIGO I-IV uterine carcinosarcoma and optimum debulking (postoperative residual tumor < 1cm) may be enrolled only if cisplatin-ifosfamide combination therapy is not feasible.
* Patients with metastatic uterine carcinosarcoma may be enrolled only if Ifosfamide/Paclitaxel combination therapy is not feasible.
* Patients with metastatic leiomyosarcoma may be enrolled only if gemcitabine-docetaxel combination therapy is not feasible.
* Measurable (target lesion) tumor, evaluable (non-target lesion) tumor or histological documentation
* No more than one prior chemotherapy. Any prior platinum or anthracycline- containing chemotherapy must have been completed more than 6 months previously
* Prior radiotherapy ≤ 25% of the hematopoietic system is allowed provided it took place more than 6 weeks before recruitment
* Patients are allowed to have received prior anticancer hormone therapy or specific immunotherapy. Patients must have completed these therapies at least three weeks before recruitment to the study
* All women with a theoretical possibility of pregnancy must produce a negative pregnancy test (serum or urinary) within seven days before starting treatment
* General health of 0 - 2 on the ECOG score
* At least 18 years of age
* Estimated life expectancy above 12 weeks
* At least 3 weeks since major surgery
* Appropriate hematologic, renal and hepatic function in accordance with the following definitions:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109 /l
* Platelets ≥ 100 × 10 9/l
* Total bilirubin ≤ 1.25 times upper limit of normal
* Estimated GFR ≥ 50 ml/min
* LVEF > 50 %
* Informed consent must be obtained from all patients.

Exclusion Criteria:

* More than one prior chemotherapy (or radiochemotherapy)
* Active infection or other serious medical impairment liable to affect the patient's ability to receive treatment according to protocol.
* Administration of other chemotherapy drugs or other anticancer hormone treatments during the study.
* History of clinically manifest atrial or ventricular arrhythmia (> LOWN II) and congestive heart failure, even if controlled by drugs (NYHA class > II). Documented myocardial infarction within 6 months before study enrollment.
* Pregnant or breastfeeding women, or women not practicing appropriate birth control methods
* Participation in another study using experimental drugs within the last 30 days
* Any other conditions or therapies which the physician believes might put the patient at risk or impair the study objective.
* Known hypersensitivity to carboplatin or pegylated liposomal doxorubicin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-06; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Anticancer activity in terms of progression-free survival time (PFS) | every 3 months

SECONDARY OUTCOMES:
Tolerability, i.e. type, frequency, severity and duration of adverse reactions (CTCAE,Version 3.0) | until recovery of toxicities
Anticancer activity in patients with measurable or evaluable disease in terms of response rates (CR, PR, SD, PD) according to RECIST criteria | six months
Overall survival | 30 months
Correlation of tumor marker CA-125 with imaging methods | six months

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Harter, MD, Principal Investigator — Klinikum Essen Mitte
Locations (15):
- Germany (15):
  - Charité, Campus Virchow Klinikum, Frauenklinik, Berlin
  - Malteser Krankenhaus, Gynäkologie und Geburtshilfe, Bonn
  - Klinikum Bremen-Mitte gGmbH, Frauenklinik, Bremen
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Frauenheilkunde und Geburtshilfe, Dresden
  - Evangelisches Krankenhaus Düsseldorf, Frauenklinik, Düsseldorf
  - Universitätsklinikum Essen, Frauenklinik, Essen
  - Klinikum der J. W. Goethe-Universität, Klinik für Gynäkologie und Geburtshilfe, Frankfurt
  - University Hospital Hamburg-Eppendorf, Hamburg
  - Gynäkologisch-onkologische Praxis, Hanover
  - St. Vincentius Kliniken AG, Frauenklinik, Karlsruhe
  - Universitätsklinikum Giessen und Marburg GmbH, Klinik für Gynäkologie, Gynäkologische Endokrinologie und Onkologie, Marburg
  - Klinikum Großhadern, Frauenklinik, München
  - Universitätsklinikum Tübingen, Frauenklinik, Tübingen
  - Universitätsklinikum Ulm, Universitätsfrauenklinik, Ulm
  - Dr. Horst Schmidt Kliniken GmbH, Klinik für Gynäkologie und gynäkologische Onkologie, Wiesbaden

IPD SHARING:
Plan to Share IPD: No